CLINICAL TRIAL: NCT03030196
Title: Denosumab and Male Infertility: a Randomized Controlled Double-blinded Intervention Study
Brief Title: Denosumab and Male Infertility: a RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01112016; 2016-003546-84 (EudraCT Number)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab (Active Comparator): subcutaneous injection with 60 mg Denosumab once
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): subcutaneous injection with NaCl once
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — NaCl 0.9% injection is used as placebo
  Other Names: Prolia

SUMMARY:
To determine the significance of systemic RANKL inhibition for male reproduction, conducting a clinical controlled randomized double blinded intervention study on infertile men, to investigating whether Denosumab (Prolia) can increase semen quality and to investigate what subgroup of infertile men that might benefit from treatment.

DETAILED DESCRIPTION:
INTRODUCTION

Infertility is a serious problem estimated to affect 7-26% of all couples globally (1;2). Approximately 9% of all newborns were conceived by assisted reproductive techniques in 2013 in Denmark (Danish Fertility Society). Impaired semen quality is the causal or contributing factor in almost 50% of all cases of infertility (3;4). Today, there exist no treatments that can improve semen quality of most infertile men. Instead, the vast majority of infertile couples are treated with assisted reproductive techniques (ART) independently of the aetiology (maternal/paternal) causing the infertility (3;5-8). The treatment choice ranges from mild intrauterine inseminations (IUI) to more invasive in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI). ART is successful for more than 70% of all couples. However, ART is very expensive and associated with maternal side effects due to the invasive methodology and the need for hormonal treatment, often for several months (9-11). Infertility is also a financial burden to society due to the costs of ART to maintain an acceptable annual birth rate.

Fertility potential determined by semen quality is established already as a fetus (12). In case the testes don't develop normally, reduced semen quality in adulthood will be the result as a result of impaired Sertoli cell function. Up until today it has barely been investigated whether intervention during adulthood can improve semen quality.

Our recent studies using both human testis and Vitamin D receptor knock-out mice revealed that the vitamin D regulated bone factor RANKL is expressed in the testis (13;14). This is a novel finding, because up until now RANKL has only been known to affect bone homeostasis and to some extend influence the immune system, inflammation and lactation (15;16). In the skeleton RANKL is expressed in osteoblasts and binds to its specific receptor RANK in osteoclasts to induce osteoclastogenesis and bone resorption (17). This activation is controlled by osteoprotegerin (OPG), which binds to the ligand domain of RANKL and thus inhibits RANK activation and osteoclastogenesis, ultimately reducing bone resorption (18). This knowledge has been utilized into development of an OPG-analogue drug, a recombinant human monoclonal IGg2 antibody Denosumab (Prolia by Amgen), which inhibits RANKL and thereby bone resorption and is indicated for use in both osteoporosis and bone metastases (19;20). Prolia has in several clinical studies shown to be safe and is approved as treatment for osteoporosis in both men and women (21-24). Newer data indicate that RANKL/OPG may be involved in regulation of pancreatic function, insulin and glucagon production which support a possible indirect effect on reproduction through bone-pancreatic-gonadal axis.

AIM OF STUDY

To determine the significance of systemic RANKL inhibition for male reproduction by investigating whether Denosumab (Prolia) can increase semen quality and particularly to identify the group of men that will benefit from the treatment.

DESIGN

Single center, prospective randomized double blinded* clinical controlled intervention.

Patients and methods:

95 infertile men, otherwise healthy, will be recruited among men referred to investigation for infertility at the outpatient clinic at Dpt. of Growth and Reproduction, Rigshopitalet. Neither choosing to participate, nor declining, will affect further outpatient clinic treatment.

The 95 participants are randomly allocated to receiving either

* Denosumab s.c. injection 60 mg x1, or
* Placebo, Sodium Chloride s.c. injection x 1

All participants deliver semen samples, blood samples and have DXA-scan performed before and after intervention. All receive supplements with Vitamin D and calcium to avoid hypocalcaemia, a known, temporary side effect to Denosumab.

*double blinded studies require that placebo and active substance are identical. Placebo can only be obtained from Amgen and we were not able to receive or purchase placebo. Instead the study will be double blinded to patient, medical doctors and all who participates in data-handling and analyses - only one nurse giving the medicine will be unblinded. She will know whether she injects active substance or placebo.

Inclusion criteria

* Men > 18 years of age referred due to infertility in need for further investigation with
* Sperm concentration ≥ 0,05 mio./ml.
* Sperm concentration <15 mio./ml or
* <40 % motile spermatozoer (ABC) or
* <4 % morphologically normal sperm (strict criteria)

Exclusion criteria

* Men with chronic diseases (diabetes mellitus, thyroid disease, endocrine diseases requiring treatment, malignant diseases or diseases known to be affected by- or interfere with vitamin D supplements (granulomatous diseases such as sarcoidosis, tuberculosis, wegeners, vasculitis as well as inflammatory bowel diseases e.g. chron's disease or ulcerative colitis etc.).
* Men with active or previous malignant disease
* Any case with indication for testis biopsy,
* Total calcium < 2.14 mmol/l
* 25-OH Vitamin D < 25 nmol/L
* Poor dental status or dental implants
* Men with obstructive oligospermia or who has been vasectomized
* Serum Inhibin B < 30 pg/ml
* Abnormal karyotype
* Patients practicing excessive exercise

SAMPLE SIZE CALCULATION AND STATISTICS

With a test level of 5% (level of significance), a power of 80% and 40 men in each group will we be able to detect a change in total number of motile sperm of 75%, and a change in sperm concentration (indexed to baseline value) of 25%.

We expect to include a total of 95 men, to take into account the possibility of dropouts. This corresponds to a dropout rate of 10%, in case the rate is lower, chances of detecting a significant difference will be above 80%.

Since we expect 50% of all infertile men in the outpatient clinic, to meet inclusion criteria and 50% of these to consent to participation, we anticipate screening of 380 men in total.

BIOSTATISTICAL ANALYSIS

All the analyses will be performed according to Good Clinical Practice guidelines and the primary analyses in the intention-to-treat population, which included all patients who underwent randomization and received the first dose of medicine on day 1. We will analyze the data in 2 ways. The primary analysis will proceed according to the randomized group assignment. The secondary analysis will be based on stratifying the men according to subgroup analyses in relation to the predefined primary and secondary endpoints.

The primary end points for this protocol will be changes in sperm production evaluated by: total motile spermatozoa (106), total progressive motile spermatozoa (106), total spermatozoa (106) or sperm concentration (106/ml). Due to the low sample size and large intraindividual variation in sperm production primary endpoints will also be evaluated after normalization to the mean average level prior to the intervention. Based on the first intervention estimated 60% of the men will benefit from the treatment and this study is designed to determine whether serum OPG, RANKL or phosphate can be used to identify men who will benefit from the treatment. The use of these specified endpoints will be useful for determining efficacy. Multiple secondary endpoints exist but for the initial investigation focus will be on: Sperm DFI, morphology, motility, semen volume, pregnancy rate, Inhibin B, vitamin D and calcium homeostasis. Subjects who terminate participation after visit at 80 days but before visit day 160 will be included for data analysis up to day 80. Men that only deliver one semen sample or have missing data at any visit will still be included in the analysis. Men with fever up to 3 months prior to semen analysis will be considered as a potential confounder. Those values will then be carried forward for analyses. A significance level of 5% is used. For the primary analyses Bonferroni-Holm p-value correction is calculated additionally. For the secondary analysis no multiple test correction are used. Instead results are discussed in view of the multiple testing situations.

1. Analyses between placebo versus active substance: The first step will be to compare the changes in primary outcomes across the two groups. This analysis will show if there is a significant difference between groups. For all endpoints measured at baseline and day 80 and 160, paired t-tests will be used to assess whether there is a significant difference between the groups and determine whether the mean change within each group differs significantly from zero. In both cases, data will be transformed as necessary to meet model assumptions. Due to assumed differences in duration of abstinence the same analyses will be conducted after exclusion of men with duration <48 hours prior to or after 80 days treatment. Afterwards, the initial analysis will be conducted by using multiple regression with relevant confounders such as season, BMI, smoking, age, duration of abstinence, time from ejaculation to motility assessment, fever etc. to see if this changes the results. For outcomes measured that cannot be compared with t-test or other parametric tests at day 1, day 80 and day 160, groups will be compared using non-parametric tests such as Wilcoxon Mann-Whitney test. For Binary outcome the data will be compared between the two groups by means of conditional logistic-regression analysis with adjustment for relevant confounders (defined as being significantly p<0.05 associated). For outcomes measured repeatedly, this will entail comparing the estimated slopes, or rates of change, of each outcome between the groups. Mixed models allow for the correlation between the repeated observations baseline-day 1-day 80- day 160 from each man to be suitably incorporated into parameter estimation. Sperm production variables will be normalized to baseline levels to avoid the huge interindividual variation in sperm count and sperm concentration
2. Subgroup analysis will be essential in this study because we expect that around 60% of the men will benefit from treatment with Denosumab. Analyses after stratification into subgroups will therefore be used to identify a marker for selecting the men who will benefit from the treatment Subjects will be grouped according to their serum OPG and/or RANKL, RANKL/OPG ratio, their DNA-fragmentation-Index prior to the start of intervention. Afterwards other potential predictors of treatment response will be tested such as BMI, S-calcium, s-phosphate, BMD, semen quality, Inhibin b, FSH at day 80 and day 160. For Serum OPG such stratification could be in two groups separated by for instance 3 pg/ml or three groups, <3, 3-4 and above 4pg/ml. Likewise for RANKL and RANKL/OPG ratio and for DNA-fragmentation-Index stratification could also be in two groups separated by e.g. DFI of 40%. The subgroup analyses will be in accordance with normal clinical practice and stratification in appropriate groups according to the clinical or highest/lowest groups.

SCREENING AND TIME COURSE

The study will be initiated January 2017 and ends when the last person has been included latest January 2021.

OUTCOME MEASUREMENTS

Endpoints:

Primary endpoints

• Change in semen production (total motile spermatozoa, progressive motile spermatozoa, sperm count, sperm concentration)

Secondary endpoints

* Change in semen quality (-motility, -morphology, semen volume)
* Change in DNA fragmentation (DFI)rate in sperm
* Change in serum Inhibin-B
* Change in serum levels of reproductive hormones (FSH, LH, AMH, testosterone, estradiol and SHBG)
* Change in serum prolactin level
* Change in fasting glucose level
* Change in fastin insulin level
* Change in c-peptide
* Change in HbA1c
* Change in lipid profile
* Change in bone mineral density evaluated by DXA.
* Change in serum level of inactive vitamin D, 1,25(OH)2D3, 25-OHD3, 24,25(OH)2D3, PTH, alkaline phosphatase, ionized calcium, phosphate, FGF23, Klotho, osteocalcin, matrix gla, osteopontin, calcitonin, pnp, procollagen III, OPG, RANKL, Sclerostin as well as other bone marker.
* Change in choice of assisted reproductive assistance technique as well as conceived pregnancies
* Change in spontaneous conception rate
* Change in live birth rate
* Change in number of spermatozoa expressing RANKL
* Change in semen pH, HCO3-, calcium, zink, phosphate, RANKL, RANK, OPG, FGF23, Klotho, osteocalcin, osteopontin. VDB, 24,25OH2
* Difference in infection rate in the two groups

SETTING, SCIENTIFIC PLAN AND RECRUITMENT

Participants will be included among men referred to the Department of Growth and Reproduction (dept. of GR), Rigshospitalet (RH) for evaluation of male infertility

This is a prospective, double blinded, two-arm randomized controlled trial. Group of intervention: Each man will receive Denosumab 60 mg x 1 sc at day 1 only Group receiving placebo: Will follow the same chain of events, although Denosumab will be replaced with saline

All men will be offered the same vitamin D and calcium supplementation starting prior to initiation of the treatment start of Denosumab or placebo: vitamin D 15 microgram and calcium 400 mg once daily.

PARTICIPANTS

Screening of ~500 infertile men will be performed. The investigators assume that ~300 men will be excluded and ~100 men do not wish to participate. Thus, 95 men will be included in the study and half will be randomized to active treatment. The investigators expect a small drop out (<5) because of high motivation and no adverse effects.

ANALYSIS AND INTERVENTION

Reproductive hormones and semen will be analyzed at dept. of GR, Rigshospitalet.

ETHICS AND SIDE EFFECTS

All the patients will have full-filled their investigation, before they are invited to the study. They will be informed of potential adverse effects, and they can leave the trial at any point without any consequences.

Denosumab is proven to be safe in several randomized studies, and is already approved by both FDA and EMA. All side effects will be closely monitored, registered and in case of either unexpected frequency of adverse effects or unexpected clinical complications it will be published.

Based on previous fertility studies at our department we expect a large proportion of the out clinic-patients will wish to participate. In our opinion the outlined study is ethical sound, and we believe that in order to generate future recommendations, randomized clinical trials are necessary.

PUBLICATION OF RESULTS

All results, positive or negative will be submitted to peer reviewed scientific journals. Data will successively be obtained and transferred to a statistical database.

ELIGIBILITY:
Inclusion Criteria:

* Men > 18 years of age refered due to infertility in need for further investigation with
* Sperm count > 0,05 mio./ml.
* The men have either sperm count <15 mio./ml or
* <40 % motile spermatozoer (A) or
* <4 % morphological normale spermatozoer (strict criteria)

Exclusion Criteria:

* Men with chronic diseases (diabetes mellitus, thyroid disease, endocrine diseases requiring treatment, malignant diseases or diseases known to be affected by- or interfere with vitamin D supplements (granulomatous diseases such as sarcoidosis, tuberculosis, wegeners, vasculitis as well as inflammatory bowel diseases e.g. chron's disease or ulcerative colitis etc).
* Men with active or previous malignant disease
* Any case with indication for tesis biopsy,
* Serum ionized calcium < 1,15 mmol/l
* Total calcium < 2.14 mmol/l
* Poor dental status og dental implants
* Men with obstructive oligospermia or who has been vasectomized
* Serum Inhibin B < 30 pg/ml
* Abnormal karyotype
* Patients practising excessive exercise

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Change in semen production (total motile spermatozoa, progressive motile spermatozoa, spermatozoa-count, spermatozoa-concentration) | 80 days and 160 days after intervention
  semen analysis

SECONDARY OUTCOMES:
Change in semen quality (-motility, -morphology of semen volume) | 80 days,160 days after intervention
  semen analysis
Change in DNA fragmentation (DFI) in spermatozoa | 80 days after intervention
  semen analysis
Change in serum Inhibin-B concentration | 80 days and 160 days after intervention
  blood sample
Change in serum levels of reproductive hormonea (FSH, LH, AMH, testosterone, estradiol inhibin B/FSh ratio and SHBG) | 80 days and 160 days after intervention
  blood sample
Change in bone mineral density evaluated by DXA | 80 days and 160 days after intervention
  DXA
• Change in serum level of inactive vitamin D, 1,25(OH)2D3, 25-OHD3, 24,25(OH)2D3, PTH, alkaline phosphatase, ionized calcium, phosphate, FGF23, Klotho, osteocalcin | 80 days and 160 days after intervention
  blood sample
Change in choice of assisted reproductive assistance technique as well as conceived pregnancies | 80 days,160 days and 365 days after intervention
  patient file
Change in spontaneous conception rate. | 80 days,160 days and 365 days after intervention
  patient file, interview
Change in number of spermatozoa expressing RANKL | 80 days and 160 days after intervention
  cytospin
Change in semen pH, HCO3-, calcium, zink, phosphate, RANKL, RANK, OPG, FGF23, Klotho, osteocalcin, osteopontin. | 80 days and 160 days after intervention
  seminal anlysis
Difference in infection rate in the two groups | 80 days and 160 days after intervention
  patient history
Change in serum level of osteopontin, calcitonin, pnp, procollagen III, OPG, RANKL, Sclerostin as well as other bone marker | 80 days and 160 days after intervention
Change in live birth rate | 80 days,160 days and 365 days after intervention
  patient file telephone interview
Change in serum prolactin level | 80 and 160 days after intervention
Change in fasting glucose level | 80 and 160 days after intervention
Change in lipid profile | 80 and 160 days after intervention
Change in fasting insulin level Change in c-peptide Change in HbA1c | 80 and 160 days after intervention
succesful fertilization (blastocyst) versus pregnancies versus live birth | 365 days after intervention
  spontaneous, IVF, ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Li J Mortensen, MD, Principal Investigator — Rigshospitalet, Dpt. of Growth and Reproduction, section GR 5064, Blegdamsvej 9, 2100 Copenhagen, Denmark; martin Blomberg Jensen, MD, Study Chair — Rigshospitalet, Dpt. of Growth and Reproduction, section GR 5064, Blegdamsvej 9, 2100 Copenhagen, Denmark
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boivin J, Bunting L, Collins JA, Nygren KG. International estimates of infertility prevalence and treatment-seeking: potential need and demand for infertility medical care. Hum Reprod. 2007 Jun;22(6):1506-12. doi: 10.1093/humrep/dem046. Epub 2007 Mar 21. PMID 17376819
- [Background] Lunenfeld B, Van Steirteghem A; Bertarelli Foundation. Infertility in the third millennium: implications for the individual, family and society: condensed meeting report from the Bertarelli Foundation's second global conference. Hum Reprod Update. 2004 Jul-Aug;10(4):317-26. doi: 10.1093/humupd/dmh028. Epub 2004 Jun 10. PMID 15192057
- [Background] Krausz C. Male infertility: pathogenesis and clinical diagnosis. Best Pract Res Clin Endocrinol Metab. 2011 Apr;25(2):271-85. doi: 10.1016/j.beem.2010.08.006. PMID 21397198
- [Background] Huynh T, Mollard R, Trounson A. Selected genetic factors associated with male infertility. Hum Reprod Update. 2002 Mar-Apr;8(2):183-98. doi: 10.1093/humupd/8.2.183. PMID 12099633
- [Background] Jain T, Gupta RS. Trends in the use of intracytoplasmic sperm injection in the United States. N Engl J Med. 2007 Jul 19;357(3):251-7. doi: 10.1056/NEJMsa070707. PMID 17634460
- [Background] Kupka MS, Ferraretti AP, de Mouzon J, Erb K, D'Hooghe T, Castilla JA, Calhaz-Jorge C, De Geyter C, Goossens V; European IVF-Monitoring Consortium, for the European Society of Human Reproduction and Embryology. Assisted reproductive technology in Europe, 2010: results generated from European registers by ESHREdagger. Hum Reprod. 2014 Oct 10;29(10):2099-113. doi: 10.1093/humrep/deu175. Epub 2014 Jul 27. PMID 25069504
- [Background] European IVF-monitoring programme (EIM) for the European Society of Human Reproduction and Embryology (ESHRE); Andersen AN, Gianaroli L, Felberbaum R, de Mouzon J, Nygren KG. Assisted reproductive technology in Europe, 2002. Results generated from European registers by ESHRE. Hum Reprod. 2006 Jul;21(7):1680-97. doi: 10.1093/humrep/del075. Epub 2006 Apr 3. PMID 16585126
- [Background] Baird DT, Collins J, Egozcue J, Evers LH, Gianaroli L, Leridon H, Sunde A, Templeton A, Van Steirteghem A, Cohen J, Crosignani PG, Devroey P, Diedrich K, Fauser BC, Fraser L, Glasier A, Liebaers I, Mautone G, Penney G, Tarlatzis B; ESHRE Capri Workshop Group. Fertility and ageing. Hum Reprod Update. 2005 May-Jun;11(3):261-76. doi: 10.1093/humupd/dmi006. Epub 2005 Apr 14. PMID 15831503
- [Background] Bhattacharya S. Effective use of assisted reproduction. Hum Fertil (Camb). 2003 May;6 Suppl 1:S60-2. doi: 10.1080/1464770312331369283. PMID 12869781
- [Background] Engel JB, Schultze-Mosgau A, Diedrich K. Five years' clinical use of GnRH antagonists: evaluation of safety and allergic potential. Reprod Biomed Online. 2005 Jun;10 Suppl 3:61-5. doi: 10.1016/s1472-6483(11)60392-1. PMID 23577417
- [Background] Engmann L, Shaker A, White E, Bekir JS, Jacobs HS, Tan SL. Local side effects of subcutaneous and intramuscular urinary gonadotropins for ovarian stimulation in in vitro fertilization: a prospective, randomized study. Fertil Steril. 1998 May;69(5):836-40. doi: 10.1016/s0015-0282(98)00043-0. PMID 9591489
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Main KM. Testicular dysgenesis syndrome: an increasingly common developmental disorder with environmental aspects. Hum Reprod. 2001 May;16(5):972-8. doi: 10.1093/humrep/16.5.972. PMID 11331648
- [Background] Blomberg Jensen M, Jorgensen A, Nielsen JE, Steinmeyer A, Leffers H, Juul A, Rajpert-De Meyts E. Vitamin D metabolism and effects on pluripotency genes and cell differentiation in testicular germ cell tumors in vitro and in vivo. Neoplasia. 2012 Oct;14(10):952-63. doi: 10.1593/neo.121164. PMID 23097629
- [Background] Jeong JH, Jin JS, Kim HN, Kang SM, Liu JC, Lengner CJ, Otto F, Mundlos S, Stein JL, van Wijnen AJ, Lian JB, Stein GS, Choi JY. Expression of Runx2 transcription factor in non-skeletal tissues, sperm and brain. J Cell Physiol. 2008 Nov;217(2):511-7. doi: 10.1002/jcp.21524. PMID 18636555
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Anastasilakis CD, Makras P. Long-term treatment of osteoporosis: safety and efficacy appraisal of denosumab. Ther Clin Risk Manag. 2012;8:295-306. doi: 10.2147/TCRM.S24239. Epub 2012 Jun 19. PMID 22767993
- [Background] Kearns AE, Khosla S, Kostenuik PJ. Receptor activator of nuclear factor kappaB ligand and osteoprotegerin regulation of bone remodeling in health and disease. Endocr Rev. 2008 Apr;29(2):155-92. doi: 10.1210/er.2007-0014. Epub 2007 Dec 5. PMID 18057140
- [Background] Khosla S. Minireview: the OPG/RANKL/RANK system. Endocrinology. 2001 Dec;142(12):5050-5. doi: 10.1210/endo.142.12.8536. PMID 11713196
- [Background] Makras P, Polyzos SA, Papatheodorou A, Kokkoris P, Chatzifotiadis D, Anastasilakis AD. Parathyroid hormone changes following denosumab treatment in postmenopausal osteoporosis. Clin Endocrinol (Oxf). 2013 Oct;79(4):499-503. doi: 10.1111/cen.12188. Epub 2013 Apr 1. PMID 23452098
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Terpos E. RANKL inhibition for the management of patients with benign metabolic bone disorders. Expert Opin Investig Drugs. 2009 Aug;18(8):1085-102. doi: 10.1517/13543780903048929. PMID 19558335
- [Background] Schwarz P, Rasmussen AQ, Kvist TM, Andersen UB, Jorgensen NR. Paget's disease of the bone after treatment with Denosumab: a case report. Bone. 2012 May;50(5):1023-5. doi: 10.1016/j.bone.2012.01.020. PMID 22586699
- [Background] Polyzos SA, Singhellakis PN, Naot D, Adamidou F, Malandrinou FC, Anastasilakis AD, Polymerou V, Kita M. Denosumab treatment for juvenile Paget's disease: results from two adult patients with osteoprotegerin deficiency ("Balkan" mutation in the TNFRSF11B gene). J Clin Endocrinol Metab. 2014 Mar;99(3):703-7. doi: 10.1210/jc.2013-3762. Epub 2014 Jan 16. PMID 24433001
- [Background] Papapoulos S, Chapurlat R, Libanati C, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Man Z, Mellstrom D, Radominski SC, Reginster JY, Resch H, Roman Ivorra JA, Roux C, Vittinghoff E, Austin M, Daizadeh N, Bradley MN, Grauer A, Cummings SR, Bone HG. Five years of denosumab exposure in women with postmenopausal osteoporosis: results from the first two years of the FREEDOM extension. J Bone Miner Res. 2012 Mar;27(3):694-701. doi: 10.1002/jbmr.1479. PMID 22113951
- [Background] Boonen S, Adachi JD, Man Z, Cummings SR, Lippuner K, Torring O, Gallagher JC, Farrerons J, Wang A, Franchimont N, San Martin J, Grauer A, McClung M. Treatment with denosumab reduces the incidence of new vertebral and hip fractures in postmenopausal women at high risk. J Clin Endocrinol Metab. 2011 Jun;96(6):1727-36. doi: 10.1210/jc.2010-2784. Epub 2011 Mar 16. PMID 21411557
- [Derived] Yahyavi SK, Holt R, Juel Mortensen L, Boisen IM, Arting LB, Jorgensen A, Juul A, Blomberg Jensen M. Effect of a single-dose denosumab on mineral homeostasis in infertile men: insights from a pilot intervention study and a randomized controlled trial. BMC Med. 2025 Mar 7;23(1):145. doi: 10.1186/s12916-025-03958-7. PMID 40055742